CLINICAL TRIAL: NCT03499574
Title: A Randomised Controlled Feasibility Trial of Dysphagia Therapy Using Biofeedback in Patients With Acute Stroke
Brief Title: Feasibility Study of Biofeedback in Dysphagia Therapy Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17028
Record Dates: First submitted 2017-11-29; First posted 2018-04-17 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Stroke, Acute; Dysphagia, Oropharyngeal
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback group (Experimental): Dysphagia therapy using surface EMG as biofeedback - 10 x 45 minute sessions of swallow strength and skill training using surface electromyography as biofeedback tool. This group will also receive usual care provided by Speech and Language Therapists, which may involve assessment, review, therapy, patient/family education.
  Interventions: Behavioral: Dysphagia therapy using surface EMG as biofeedback; Behavioral: Usual Care
- Control group (Other): This group will receive usual care provided by Speech and Language Therapists, which may involve assessment, review, therapy, patient/family education
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Dysphagia therapy using surface EMG as biofeedback — 10 x 45 minute sessions over 14 days
  Other Names: Biofeedback
  Arms: Biofeedback group
Behavioral: Usual Care — Usual care may include the following Speech and Language Therapy interventions; assessment, review, therapy, patient/family education etc.. Dose will vary.

SUMMARY:
This study will investigate the feasibility of delivering swallowing therapy using surface electromyography as a means of biofeedback to patients with dysphagia in the acute stroke setting. It will investigate trends in efficacy by comparing biofeedback therapy to usual care. The results will inform future dosing and efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis stroke, new dysphagia, medically stable, adequate trunk strength for videofluoroscopy.

Exclusion Criteria:

* Severe cognitive impairment, previous dysphagia, previous neurological condition, severe visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | 2 weeks
  Count of number of participants can be recruited
Number of participants completing the treatment | 2 weeks
  Count of number of participants completing the treatment
Average number of sessions completed | 2 weeks
  Average number of sessions completed across participants.

SECONDARY OUTCOMES:
Change in Swallow function - severity | Pre and post 3 week intervention intervention and at 90 days
  Using Dysphagia Severity Rating Scale - scale of 0-16. 0 is normal, 16 is the most severe.
Change in Swallow function - intake | Pre and post 3 week intervention intervention and at 90 days
  Functional Oral Intake Scale - 7 point scale from 1-7. Higher number indicated increased amount and normality of oral intake.
Change in Swallow physiology - PAS | Pre and post 2 week intervention
  Videofluoroscopy assessment to measure swallow safety with regards to penetration/aspiration using the Penetration Aspiration Scale (PAS). 8 point scale. The higher the number the increase in penetration/aspiration.
Change in swallow physiology - timing | Pre and post 2 week intervention
  Videofluoroscopy assessment to measure timing of swallow physiology
Quality of life | Pre and post 2 week intervention and at 90 days
  Dysphagia Handicap Index
Change in Clinical outcomes - disability | Pre and post 2 week intervention and at 90 days.
  Disability - using the Modified Rankin scale. Scale from 0-6 with higher numbers signifying increased disability
Change in Clinical outcomes - stroke severity | Pre and post 2 week intervention
  Stroke severity - NIHSS. Scale from 0-42. Increased number means increase in stroke severity.
Change in Clinical outcomes - tube status | Pre and post 2 week intervention and at 90 days.
  Feeding tube status
Change in Clinical outcomes - mortality | Pre and post 2 week intervention and at 90 days.
  Mortality
Change in Clinical outcomes - pneumonia | Pre and post 2 week intervention and at 90 days.
  Presence of pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Timothy England, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No